CLINICAL TRIAL: NCT02146157
Title: A Randomized, Double-blind, Placebo-controlled Trial to Assess Efficacy and Tolerability of an Herb and Mineral Combination Product on Fasting Glucose in Adults at Risk for Developing Diabetes
Brief Title: Trial of an Herb and Mineral Combination Product on Fasting Glucose in Adults at Risk for Developing Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NewChapter, Inc. (Industry)
Collaborators: Procter and Gamble (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 2012110
Record Dates: First submitted 2014-04-07; First posted 2014-05-23 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2015-10

CONDITIONS: Prediabetes
MeSH Terms: conditions — Prediabetic State

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- herb and mineral combination product (Active Comparator): Subjects will consume 3 herb and mineral combination product softgels daily, 1 softgel immediately before each of the 3 largest meals, throughout the 12-week supplementation period.
  Interventions: Dietary Supplement: herb and mineral combination product
- placebo (Placebo Comparator): Subjects will consume 3 softgels daily, 1 softgel immediately before each of the 3 largest meals, throughout the 12-week supplementation period
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: herb and mineral combination product — herb and mineral product containing cinnamon, turmeric and holy basil
  Arms: herb and mineral combination product
Dietary Supplement: Placebo — Placebo of herb and mineral product containing cinnamon, turmeric and holy basil
  Arms: placebo

SUMMARY:
This is a multi-center, randomized, double-blind, placebo-controlled study in approximately 104 subjects (52 per group) to evaluate the effectiveness of an herb and mineral combination product on fasting serum glucose levels in subjects with impaired fasting glucose. The study consists of 5 visits: a Screening visit, followed by a Baseline visit (at which eligible subjects will be randomized to product to consume throughout the 12-week supplementation period), followed by Supplementation period visits at 3, 6 and 12 weeks after baseline.

DETAILED DESCRIPTION:
The target population of this clinical trial is otherwise healthy, pre-diabetic adults who present with impaired fasting glucose.

ELIGIBILITY:
Inclusion Criteria:

* Be male or female, at least 18 years of age
* If age ≥45 years, must have a body mass index ≥ 25 kg/m2
* If age <45 years, must have a body mass index ≥ 25 kg/m2 AND present with at least one additional risk factors for developing diabetes.
* Agree to use contraception throughout study period, unless postmenopausal or surgically sterile (women only)
* Be able to understand the nature and purpose of the study including potential risks and side effects
* Be willing to consent to study participation and to comply with study requirements
* Have a finger stick fasting blood glucose between 105 and 140 mg/dL and a serum fasting glucose between 100 and 125 mg/dL, measured at screening

Exclusion Criteria:

* Have diabetes (type I or II) or an HBA1c measurement >6.5% at any time in the past or at the screening visit
* Have been taking within 2 weeks of screening any dietary supplement including vitamin and mineral complexes; herbal supplements; fish oil; fiber supplements; or any herbal ingredient/product that significantly affects glucose metabolism
* Have been taking within 4 weeks of screening any prescription or over-the-counter (OTC) medication that significantly affects glucose metabolism, including but not limited to, sulfonylureas, meglitinides, biguanides, thiazolidinediones, alpha-glucosidase inhibitors, Inhibitors of dipeptidyl peptidase 4 (DPP-4 inhibitors), systemic corticosteroids
* Daily use of non-steroidal anti-inflammatory drugs (NSAIDS) (daily baby aspirin use and continuous use of NSAIDS for 3 days or less for acute aches and pains are acceptable)
* Any co-morbidity or treatment that could, in the opinion of the investigator, preclude the subject's ability to successfully and safely complete the study or that may confound study outcomes
* Anticipated changes in dietary patterns or physical activity levels during the study, including attempts at body weight reduction
* Eating disorder
* Polycystic ovary syndrome
* Known allergies or intolerance to any substance in the study product
* Are pregnant or breastfeeding women
* History of alcohol, drug, or medication abuse
* Have participated in another study with any investigational product within 1 month of screening
* Had a recent (<3 months) gastrointestinal surgery or any planned surgery during the clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2013-02; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in fasting blood glucose | Day 84
  Fasting glucose will be measured on serum samples obtained at screening (to be used as baseline value) and at day 84

SECONDARY OUTCOMES:
Change from Baseline in fasting serum glucose | Day 42
  Fasting glucose will be measured on serum samples obtained at screening (to be used as baseline value) and at day 42
Change from Baseline in fasting blood glucose | Day 21
  Fasting glucose will be measured on serum samples obtained at screening (to be used as baseline value) and at day 21
Change from Baseline in HbA1c | Day 84
  Glycosylated hemoglobin (HbA1c) will be measured on whole blood samples obtained at screening and at day 84.
Change from Baseline in fasting lipids | Day 84
  Total cholesterol, high-density lipoprotein, low-density lipoprotein, very low-density lipoprotein, and triglycerides will be measured on serum samples obtained at screening and at day 84 using a standard lipid panel.
Change from Baseline in fasting lipids | Day 42
  Total cholesterol, high-density lipoprotein, low-density lipoprotein, very low-density lipoprotein, and triglycerides will be measured on serum samples obtained at screening and at day 42 using a standard lipid panel.
Change from Baseline in fasting lipids | Day 21
  Total cholesterol, high-density lipoprotein, low-density lipoprotein, very low-density lipoprotein, and triglycerides will be measured on serum samples obtained at screening and at day 21 using a standard lipid panel.
Change from Baseline in BMI | Day 84
  Body mass index
Change from Baseline in waist-to-hip ratio | Day 84

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Radiant Research, Chicago, Illinois
  - Central Kentucky Research Associates, Lexington, Kentucky
  - Quest Research Institute, Bingham Farms, Michigan
  - Radiant Research, Cincinnati, Ohio
  - Providence Health Partners Center for Clinical Research, Dayton, Ohio
  - Mountain View Clinical Research, Greer, South Carolina